CLINICAL TRIAL: NCT02129920
Title: Recurrent Embolism Lessened by Rivaroxaban, an Anti-Xa Agent of Early Dosing for Acute Ischemic Stroke and Transient Ischemic Attack With Atrial Fibrillation Study (RELAXED)
Brief Title: RELAXED: Recurrent Embolism Lessened by Rivaroxaban for Acute Ischemic Stroke
Acronym: RELAXED
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Japan Cardiovascular Research Foundation (Other)
Responsible Party: Principal Investigator, Kazuo Minematsu, M.D., Japan Cardiovascular Research Foundation
Other Study IDs: M25-113
Record Dates: First submitted 2014-05-01; First posted 2014-05-02 (Estimated); Last update posted 2014-05-02 (Estimated); Status verified 2014-04

CONDITIONS: Stroke, Acute; Atrial Fibrillation
Keywords: Stroke; Cerebral Infarction; Atrial Fibrillation; Arrhythmias, Cardiac; Heart Diseases; Cardiovascular Diseases; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Vascular Diseases; Brain Infarction; Brain Ischemia; Anticoagulants; Hematologic Agents; Therapeutic Uses
MeSH Terms: conditions — Stroke; Atrial Fibrillation; Cerebral Infarction; Arrhythmias, Cardiac; Heart Diseases; Cardiovascular Diseases; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Vascular Diseases; Brain Infarction; Brain Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- NVAF, acute ischemic stroke/TIA: Consecutive acute ischemic stroke/TIA patients with nonvalvular atrial fibrillation and treated with rivaroxaban
  Interventions: Other: This is an observational study

INTERVENTIONS:
Other: This is an observational study
  Other Names: This is an observational, not intervention, study.

SUMMARY:
Early recurrence of cardioembolic stroke in patients with atrial fibrillation is common, reaching approximately 6% within 30 days after initial stroke. Therefore, it is preferable to provide early anticoagulation for cardioembolic stroke. However, early anticoagulation may increase the risk of hemorrhagic transformation of cerebral infarcts. It is difficult to decide the timing of initiation for anticoagulant therapy in stroke patients with non-valvular atrial fibrillation (NVAF). In 2013 the European Heart Rhythm Association presented the practical guides for oral anticoagulants in NVAF patients, which recommend that the optimal time to start anticoagulant therapy should be determined according to the stroke severity. However, this recommendation is principally an experts' opinion and is not suitable in the clinical practice in Japan.

RELAXED, a multicenter observational study is planned to evaluate the efficacy and safety of an oral direct activated coagulation factor Xa inhibitor, rivaroxaban, for acute ischemic stroke patients with NVAF in consideration of the infarct size, timing of initiation for rivaroxaban medication, and other patient characteristics, and thereby to determine the optimal timing of the initiation during acute ischemic stroke. The consecutive acute ischemic stroke / transient ischemic attack (TIA) patients with NVAF who are treated with rivaroxaban will be enrolled. The infarction size at 0-48 hours after stroke onset will be measured by the diffusion weighted image (DWI) MRI. The primary efficacy endpoint is recurrent ischemic stroke within 3 months. The primary safety endpoint is major bleedings within 3 months. The optimal timing to initiate rivaroxaban during acute ischemic stroke is determined by analysis of co-relation between primary endpoints and the infarct size / time to initiate rivaroxaban.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of acute ischemic stroke or transient ischemic attack (TIA)
* Having non-valvular atrial fibrillation
* Visiting the clinic/hospital within 48 hours of the onset of acute ischemic stroke or TIA
* Identification of an infarct in the middle cerebral artery (MCA) territory (symptoms ascribable to ischemia in the MCA territory in TIA patients)
* Initiation of treatment with rivaroxaban within 30 days of the onset of acute ischemic stroke or TIA
* Written informed consent by patients

Exclusion Criteria:

* hypersensitivity to rivaroxaban 2) Active bleeding (clinically significant hemorrhage) including gastrointestinal hemorrhage
* liver disease complicated with coagulation disorder
* liver disorder corresponding to Child-Pugh Class B or C
* renal failure (creatinine clearance: <15 mL/minute)
* poorly controlled hypertension (higher than 180/100)
* Woman who are or are likely to be pregnant
* Ongoing treatment with HIV protease inhibitors including ritonavir, atazanavir and indinavir
* Ongoing treatment with itraconazole, voriconazole and ketoconazole
* Active bacterial endocarditis
* Patients considered by the investigator to be unsuitable for participating in this study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive acute ischemic stroke/TIA patients with nonvalvular atrial fibrillation and treated with rivaroxaban
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2014-02; Primary Completion 2016-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Recurrent ischemic stroke and major bleeding | 3 monhths
  The optimal timing to start treatment with rivaroxaban of the initiation for during acute ischemic stroke are determined by analysis of co-relation between primary endpoints including recurrent ischemic stroke / major bleeding, and the cerebral infarction size / time to start treatment with rivaroxaban.
  Major bleeding according to the criteria by the International Society of Thrombosis and Haemostasis (ISTH)

SECONDARY OUTCOMES:
ischemic stroke and transient ischemic attack | 3 months
Composite cardiovascular events | 3 months
  The composite cardiovascular events are included ischemic stroke, TIA, systemic embolism, acute coronary syndrome, deep vein thrombosis, pulmonary embolism, other ischemic disease, revascularization, total death, cardiovascular death
Any bleeding events | 3 months
Intracranial hemorrhage | 3 months
Hemorrhagic transformation of cerebral infarcts | 3 months
Adverse event | 3 month
Recurrence of ischemic stroke and major bleeding according to whether or not heparin is administered | 3 months
Recurrence of ischemic stroke and major bleeding according to whether rivaroxaban is administered in the morning or evening | 3 month
Duration of hospitalization | 3 month
Safety and efficacy of rivaroxaban administration via tube or by crush tablet | 3 month
Definite clinical data on patients developing recurrent ischemic stroke or intracranial hemorrhage during rivaroxaban medication | 3 month
Medical expenditures using a model | 3 month

CONTACTS AND LOCATIONS:
Overall Officials: Kazuo Minematsu, M.D., Principal Investigator — Japan Cardiovascular Research Foundation, and National Cerebral and Cardiovascular Center
Locations (1):
- Japan Cardiovascular Research Foundation, Suita, Osaka, Japan

REFERENCES:
- [Derived] Koge J, Yamagami H, Toyoda K, Yasaka M, Hirano T, Hamasaki T, Nagao T, Yoshimura S, Fujishige M, Tempaku A, Uchiyama S, Mori E, Koga M, Minematsu K. Early initiation of rivaroxaban after reperfusion therapy for stroke patients with nonvalvular atrial fibrillation. PLoS One. 2022 Apr 6;17(4):e0264760. doi: 10.1371/journal.pone.0264760. eCollection 2022. PMID 35385480
- [Derived] Yasaka M, Minematsu K, Toyoda K, Yamagami H, Yoshimura S, Nagao T, Mori E, Hirano T, Hamasaki T, Yamaguchi T. Design and Rationale of the RELAXED (Recurrent Embolism Lessened by rivaroxaban, an Anti-Xa agent, of Early Dosing for acute ischemic stroke and transient ischemic attack with atrial fibrillation) Study. J Stroke Cerebrovasc Dis. 2016 Jun;25(6):1342-8. doi: 10.1016/j.jstrokecerebrovasdis.2016.01.035. Epub 2016 Mar 14. PMID 26987488